CLINICAL TRIAL: NCT05849168
Title: High-Intensity Interval Training (HIIT) to Improve Symptoms of Deployment-Related Respiratory Disease - A Pilot Study
Brief Title: High-Intensity Interval Training to Improve Symptoms of Deployment-Related Respiratory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2069
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Occupational Exposure
Keywords: exercise tolerance; exercise therapy; airborne hazards; deployment-related respiratory disease; veterans; burn pit
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Veterans with respiratory symptoms (Experimental)
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Participants will complete a 12-week exercise training program. The program consists of 3x/week HIIT sessions on an upright stationary bicycle (~40 minutes each) and 3x/week home aerobic sessions (any type of aerobic exercise; 45 minutes each).

SUMMARY:
Some military personnel who have been exposed to burn pit emissions, desert dust, and other airborne hazards experience new respiratory symptoms after deployment. The goal of this clinical trial is to learn about exercise in veterans with new respiratory symptoms after deployment to Southwest Asia. The main questions it aims to answer are:

1. Do veterans with new respiratory symptoms after deployment have heart or lung abnormalities that contribute to difficulty exercising?
2. Does high-intensity interval training (HIIT) improve fitness and symptoms?

Study participants will complete the following:

1. Study Visits 1A and 1B: Exercise test (VO2max test), echocardiogram (heart ultrasound), blood tests, questionnaires
2. Exercise program: 12 weeks of 3x/week supervised HIIT on upright stationary bicycle (~40 minutes each) and 3x/week home aerobic exercise (45 minutes each)
3. Study Visits 2A and 2B: Exercise test (VO2max test), echocardiogram (heart ultrasound), blood tests, questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Deployment of ≥30 days to Iraq, Afghanistan, Kuwait, Saudi Arabia, Bahrain, Qatar, United Arab Emirates, Kyrgyzstan, or Djibouti after September 2001
* New onset of cough, shortness of breath, chest tightness/wheezing, dyspnea on exertion or exercise intolerance which started during or after deployment
* Definite or probable distal lung disease (≥1 hyperinflation, emphysema, bronchiolitis, small airways inflammation, peribronchiolar fibrosis, or granulomatous pneumonitis on surgical lung biopsy; or ≥2 centrilobular nodularity, air trapping, mosaicism, or bronchial wall thickening on chest computed tomography [CT]), definite or probable deployment-related asthma (≥1 increase in post-bronchodilator forced expiratory volume in 1 second [FEV1] ≥12% and ≥200cc, or methacholine challenge with provocation concentration causing a 20% decline in FEV1 [PC20] ≤16 mg/mL), or unexplained dyspnea on exertion or exercise intolerance despite noninvasive testing including pulmonary function testing, methacholine challenge, transthoracic echocardiography, and/or chest computed tomography
* Current symptoms of dyspnea on exertion or exercise intolerance
* Residence <90 miles from Rocky Mountain Regional VA and ability / willingness to attend in-person HIIT sessions and research visits
* Vaccinated against Coronavirus-19 including primary series and (if eligible) ≥1 booster

Exclusion Criteria:

* Active / uncontrolled cardiovascular or pulmonary disease (e.g. hypertension with blood pressure >160/100 despite antihypertensive therapy, known hypertensive response to exercise [systolic blood pressure >220 mmHg in men / >190 mmHg in women], coronary artery disease, left ventricular ejection fraction ≤45% or heart failure with preserved ejection fraction with ongoing symptoms despite diuretic therapy, uncontrolled arrhythmia, moderate or severe valvular abnormality, diabetes with HbA1c >8.5%, asthma exacerbation requiring steroids within 4 weeks of enrollment, interstitial lung disease, untreated severe obstructive sleep apnea)
* Pre-deployment history of cardiovascular or pulmonary disease including coronary artery disease, left ventricular ejection fraction ≤45% or heart failure with preserved ejection fraction requiring diuretic therapy, arrhythmia, valvular abnormality, chronic obstructive pulmonary disease, asthma (excluding childhood asthma that did not persist into adulthood), interstitial lung disease, or pulmonary hypertension
* Body mass index <18.5 or >45
* Anemia with hemoglobin <10 g/dl
* Disorders that adversely influence exercise ability (e.g. arthritis or peripheral vascular disease)
* Current fitness program (e.g. >30 minutes at metabolic equivalents [METs] >6 3 times/week or more)
* Pregnancy or possible anticipated pregnancy during study duration
* Post-menopausal status in women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Cornwell, MD, MSCS, Principal Investigator — University of Colorado, Denver; Lindsay Forbes, MD, Principal Investigator — University of Colorado, Denver; Silpa Krefft, MD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - VA Eastern Colorado Health Care System, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Veterans With Respiratory Symptoms: Veterans with respiratory symptoms meeting the inclusion and exclusion criteria
Period: Overall Study
Arm/Group | Veterans With Respiratory Symptoms
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Oxygen Consumption (VO2max)
Description: Obtained via metabolic cart during maximal cardiopulmonary exercise testing, in ml/kg/min
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: ml/kg/min
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 12
ml/kg/min | 26.4 [23.8 to 28.9]

2. Primary Outcome: Health-related Quality of Life by Short Form 36 (SF-36) Questionnaire
Description: Units, Range 0-100 with higher scores indicating more favorable health state
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: Units on a scale, Range 0-100
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 12
Units on a scale, Range 0-100 | 67 [44 to 79]

3. Secondary Outcome: Left Ventricular Ejection Fraction Measured by Transthoracic Echocardiogram
Description: %
Time Frame: Up to 1 hour
Population: Two participants were unable to complete transthoracic echocardiography due to scheduling constraints
Measure: Median (Inter-Quartile Range); unit: % of blood
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 10
% of blood | 60 [58 to 63]

4. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion Measured by Transthoracic Echocardiogram
Description: mm
Time Frame: Up to 1 hour
Population: Two participants were unable to complete transthoracic echocardiography due to scheduling constraints
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 10
mm | 26 [21 to 29]

5. Secondary Outcome: Plasma Acylcarnitine 10:0 Measured by Peripheral Venous Metabolomics (Ultra-high Performance Liquid Chromatography Coupled to Mass Spectrometry)
Description: Relative ion count
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: Relative ion count
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 12
Relative ion count | 4448588 [3488443 to 7035835]

6. Secondary Outcome: Feasibility of Exercise Program, Reported by Participant and Measured by Responses to Questionnaire
Description: Score, Likert scale indicating agreement with the statement "I was able to complete the scheduled high-intensity interval training sessions," 5-point range from 1 = "Strongly disagree" to 5 = "Strongly agree" with "Strongly agree" indicating greater agreement
Time Frame: Up to 1 hour
Population: One participant withdrew from study
Measure: Median (Inter-Quartile Range); unit: Scores on a Likert scale, 5-point range
Arm/Group | Veterans With Respiratory Symptoms
Number analyzed (Participants) | 11
Scores on a Likert scale, 5-point range | 5 [4 to 5]

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 4 months
Arm/Group | Veterans With Respiratory Symptoms
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05849168/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05849168/ICF_001.pdf